CLINICAL TRIAL: NCT04040465
Title: Asprin Dosing Estimator in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, mark munger, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00117303
Record Dates: First submitted 2019-07-22; First posted 2019-07-31 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2020-10

CONDITIONS: Aspirin Sensitivity
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: We will place patients into 3 different groups based on BMI, and within those groups patients will be randomly assigned to an aspirin dose (81mg, 325mg, or 500mg)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Normal Weight/Low Dose Aspirin (Active Comparator): BMI 22-25 kg/m^2 & receiving 81mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Normal Weight/Normal Dose Aspirin (Active Comparator): BMI 25-30 kg/m^2 & receiving 325mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Normal Weight/High Dose Aspirin (Active Comparator): BMI > 30 kg/m^2 & receiving 500mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Overweight/Low Dose Aspirin (Active Comparator): BMI 22-25 kg/m^2 & receiving 81mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Overweight/Normal Dose Aspirin (Active Comparator): BMI 25-30 kg/m^2 & receiving 325mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Overweight/High Dose Aspirin (Active Comparator): BMI > 30 kg/m^2 & receiving 500mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Obese/Low Dose Aspirin (Active Comparator): BMI 22-25 kg/m^2 & receiving 81mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Obese/Normal Dose Aspirin (Active Comparator): BMI 25-30 kg/m^2 & receiving 325mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin
- Obese/High Dose Aspirin (Active Comparator): BMI > 30 kg/m^2 & receiving 500mg Aspirin daily for 2 weeks
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Participants will be categorized into 3 BMI groups and will be randomly given various doses of aspirin to compare effectiveness and create a dosing regimen.

SUMMARY:
Understanding sources of variability in human drug dosing is important to the beneficial and safe use of any drug. Understanding and applying the science of individualizing a drug dose to a patient is called precision medicine.

Aspirin is one of the oldest most utilized medications for its ability to lower fever, relieve pain, and to reduce the stickiness of platelets (tiny blood cells that help your body form clots to stop bleeding. Aspirin dosing is currently the same for all patients and is not individualized. In the last century, aspirin has shown benefit in reducing cancer, stroke, and preventing cardiovascular events after one has already had a heart attack or stroke. Previous human studies have not found consistent positive effects of aspirin when dosed by body weight. Therefore, how should aspirin be dosed in 2019? Aspirin resistance is the failure of aspirin to reduce platelet stickiness and thin the blood and most importantly, is associated with higher risk of heart attacks and strokes. Aspirin resistance may occur due to not taking aspirin on a regular basis, differences in how platelets behave in some persons, use of over the counter pain medicines like Motrin®, reduced amount of drug in the body, and/or a lack of being able to predict a dose for a certain individual.

To find out the best way to dose aspirin, the investigators propose to study healthy volunteers (persons without any known disease) with different ages and body sizes to see if aspirin blood levels are tied to platelet stickiness. This information will be used to mathematically build a computer-based picture of aspirin dosing that will help physicians pick the best dose of aspirin for each patient. The investigators will then extend studies for the aspirin dose estimator to be used in other countries in people with heart problems and stroke, recording future events in a randomized (i.e., coin toss) manner, to determine if the ability of the aspirin dose estimator to prevent future heart attacks and stroke compared to people receiving aspirin doses that were chosen without the estimator.

DETAILED DESCRIPTION:
AIM 1: Determine urine TXB2, platelet aggregation function testing (VerifyNow® ASA Test), salicylate level, CBC with differential, and hs-CRP, in 18 healthy volunteers across BMI classes of 22-25 (Normal Weight), >25-30 (Overweight), and > 30 kg/m2 (Obese).Total enrolled cohort: 60 patients and planned treatment cohort: 54 completed patients (anticipated dropout rate of 10% = 6 patients). The investigators have powered this sample size based on estimates of effect sizes from published studies examining platelet activation in patients across a range of BMIs and assuming an alpha = 0.05, with 80% power. In addition, height and weight as predictors will be evaluated independently of BMI. BMI patient groups (22-25, >25-30, and > 30 kg/m2) will be randomized to low-dose ASA (81mg standard-release), moderate dose ASA (325mg) or high dose ASA (500mg) (6 patients/each dose).

All patients will have a CBC with differential (to measure blood cell counts including platelets) and hs-CRP at baseline, serial urine TXB2 (-1, and 2 and 5 hours post ASA dose), platelet aggregation function testing using VerifyNow® ASA Test 15 min post ASA dose, serial salicylate levels (0, 15", 2 hours post-ASA dose) and again 10-14 days after chronic dosing (urine TXB2 2 hours post ASA dose and platelet aggregation function testing using VerifyNow® Test 15 min post ASA dose only).

AIM 2: Model associations between construct variables (BMI and aspirin dose) with predictive variables as collected in AIM 1. Multiple and Linear Regression with backward selection will be used. In addition, a Structured Equation Model will be applied to the data. Statistical assessment of model fit will be conducted for all models.

AIM 3: Build an Aspirin Dose Estimator to predict aspirin dosing. Model associations from AIM 2 will create demand estimates that will feed into a user-friendly aspirin dosage estimator. The simulator will comprise: 1) Entry: An entry screen. In this screen the user will enter the features of patient clinical information attributes. The user then clicks a 'run' button. 2) Demand Output: The simulator will then create an output screen that will show graphically aspirin dosing options.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55 years old (male or female)
* Healthy Volunteers (medication free without acute or chronic significant health problems or pathologies)

Exclusion Criteria:

* History of asthma
* History of chronic bronchitis
* History of emphysema
* History of renal impairment (eGFR < 30 ml/min)
* History of hypertension (reviewed by study staff)
* History of hyperlipidemia
* History of diabetes
* History of smoking (within last month)
* Current depression or anxiety requiring medication therapy
* Inability to finish the study for any reason
* Any current pathological condition outside of normal range
* Thrombocytopenia (platelet count < 150 K/µL)
* Other known platelet disorders (eg. von Willebrand disease, Glanzmann thrombasthenia, Bernard-Soulier Syndrome)
* Current use of dipyradamole, PGY 12 inhibitors, NSAIDs
* Or as otherwise determined by the investigative team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Height | 2 weeks per participant
  Used to measure BMI
Weight | 2 weeks per participant
  Used to measure BMI
Urine TBX2 Collection (Thromboxane levels) | 2 weeks per participant
  Thromboxane levels measured for indicator of platelet aggregation function
Salicylate Levels | 2 weeks per participant
  Used to measure amount of systemic aspirin to compare with TBX2 and BMI categories
Aspirin Reaction Units (ARU) | 2 weeks per participant
  Number given from Verifynow device that will be used to determine platelet aggregation function by arachidonic acid induced aggregation

SECONDARY OUTCOMES:
Complete Blood Count (CBC) | 2 weeks per participant
  Safety measure labs taken on 2 visits
High-sensitivity C-reactive protein (hs-CRP) | 2 weeks per participant
  Measured as an inflammatory marker and indicator of cardiac risk and risk of stroke
Blood Pressure (mmHg) | 2 weeks per participant
  Safety measure taken on 2 visits
Heart Rate (BPM) | 2 weeks per participant
  Safety measure taken on 2 visits
Respiratory Rate (breaths per minute) | 2 weeks per participant
  Safety measure taken on 2 visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No